CLINICAL TRIAL: NCT02146794
Title: Renal Denervation in Chronic Heart Failure
Acronym: REACH
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ICCH-10/065
Record Dates: First submitted 2014-05-19; First posted 2014-05-26 (Estimated); Last update posted 2014-05-26 (Estimated); Status verified 2014-05

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Renal denervation (Experimental): renal denervation
  Interventions: Device: Renal denervation

INTERVENTIONS:
Device: Renal denervation — Renal denervation
  Other Names: Symplicity Renal Denervation System

SUMMARY:
Renal denervation can be carried out for heart failure

DETAILED DESCRIPTION:
There are theoretical reasons why renal denervation might be beneficial for patients with chronic heart failure. It is not known whether they would suffer large drops in blood pressure which might compromise safety.

This pilot study required patients to remain in hospital for one week during which they had careful monitoring of blood pressure with the ability to halt the trial if any patient suffered any dangerous effect such as a large drop in blood pressure. It also monitored blood pressure after discharge for six months.

ELIGIBILITY:
Inclusion Criteria:

-Patients were required to have chronic symptomatic systolic heart failure (NYHA class III or IV) on maximal tolerated medical therapy, including beta-blocker, ACE inhibitor or angiotensin receptor blocker, and spironolactone.

Exclusion Criteria:

* Clinically unstable patients or those with significant valvular disease
* An estimated glomerular filtration rate <35 ml/min
* Unfavourable renal anatomy
* Tortuous femoral arteries were not eligible

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2011-05; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 6 months
  Renal denervation had been reported to cause a 30 mmHg fall in blood pressure when used in hypertension. Although in principle renal denervation might be favourable for physiology in chronic heart failure, numerous theoretical possibilities exist for the procedure causing deterioration in clinical status, including the possibility of a large fall in blood pressure.
  A deterioration in symptomatic status or occurrence of an event such as presyncope or syncope would be considered a primary outcome event.

SECONDARY OUTCOMES:
Systolic blood pressure | 6 months
  Monitored as inpatient for 5 days, then as outpatient for 6 months
Serum Creatinine | 6 months
Serum sodium | 6 months
Serum potassium | 6 months
6 minute walk distance | 6 months

OTHER OUTCOMES:
Left ventricular ejection fraction by Echocardiography | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Darrel P Francis, MD, Study Chair — Imperial College London; Justin E Davies, MD, Principal Investigator — Imperial College London

REFERENCES:
- [Background] Shun-Shin MJ, Howard JP, Francis DP. Removing the hype from hypertension. BMJ. 2014 Mar 6;348:g1937. doi: 10.1136/bmj.g1937. No abstract available. PMID 24603957
- [Background] Howard JP, Cole GD, Sievert H, Bhatt DL, Papademetriou V, Kandzari DE, Davies JE, Francis DP. Unintentional overestimation of an expected antihypertensive effect in drug and device trials: mechanisms and solutions. Int J Cardiol. 2014 Mar 1;172(1):29-35. doi: 10.1016/j.ijcard.2013.12.183. Epub 2014 Jan 8. PMID 24480181
- [Result] Davies JE, Manisty CH, Petraco R, Barron AJ, Unsworth B, Mayet J, Hamady M, Hughes AD, Sever PS, Sobotka PA, Francis DP. First-in-man safety evaluation of renal denervation for chronic systolic heart failure: primary outcome from REACH-Pilot study. Int J Cardiol. 2013 Jan 20;162(3):189-92. doi: 10.1016/j.ijcard.2012.09.019. Epub 2012 Sep 29. PMID 23031283